CLINICAL TRIAL: NCT05071976
Title: Near-infrared FluORescencE Assessment of Myocutaneous Flap Microperfusion for Gynecologic RecONstrucTion (FOREFRONT): A Pilot Study
Brief Title: A Study of Near-Infrared Fluorescence Imaging With ICG During Reconstructive Gynecologic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-349
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Gynecologic Surgery
Keywords: gynecologic surgery; abdominal wall reconstruction procedure; pelvic reconstruction procedure; Near-Infrared Fluorescence Imaging; ICG; 21-349; Memorial Sloan Kettering Cancer Center

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants undergoing a pelvic or abdominal wall reconstruction procedure (Experimental): Women undergoing a pelvic or abdominal wall reconstruction procedure after radical gynecologic surgery for any indication at Memorial Sloan Kettering Cancer Center
  Interventions: Diagnostic Test: ICG-NIR angiography

INTERVENTIONS:
Diagnostic Test: ICG-NIR angiography — Capture NIR video of flap site beginning at time of ICG injection. At time of subjective peak intensity, capture video of flap and recipient wound bed. Measure rate of ICG egress from the global flap at 60, 120, and 180 seconds after initial dye injection from intraoperative video

SUMMARY:
The objective of this study is to assess whether Near-Infrared Fluorescence/NIR Imaging perfusion alters intraoperative management of the flap or of the participant wound bed.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a pelvic reconstruction procedure after radical gynecologic surgery for any indication at MSK.
* Age ≥18 years.

Exclusion Criteria:

* Women with hepatic dysfunction as evidenced by elevated transaminases (two times the upper limit of normal).
* Women with a history of cirrhosis or other chronic liver disease.
* Women with a documented severe or life threatening allergy to iodine.
* Women with an allergy to ICG or severe allergy to iodinated contrast.
* Women undergoing any free flap (non-pedicled) reconstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2026-10-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases in which intraoperative ICG-NIR angiography altered surgical flap reconstruction plans | Up to 24 months
  The primary purpose of this study is to introduce ICG-NIR angiography in abdominopelvic skin and myocutaneous pedicle flap-based reconstruction during gynecologic oncology surgery and determine the percentage of cases in which intraoperative ICG-NIR angiography altered surgical flap reconstruction plans.

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Abu-Rustum, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and Followup), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Followup), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Followup), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent and Followup), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Followup), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Followup), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskc.org